CLINICAL TRIAL: NCT03415815
Title: A Real-world Observational Study to Evaluate Lymph Metastases and Prognoses of the Chinese Patients With Thoracic T1-T3 Esophageal Cancer
Brief Title: An Observational Study to Evaluate Lymph Metastases and Prognoses of the Patients With Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Yin Li, Professor, Henan Cancer Hospital
Other Study IDs: HenanEC
Record Dates: First submitted 2018-01-11; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer
Keywords: Chinese, real-world evidences, T1-T3 esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T1-T3 esophageal cancer: Pathologically diagnosed patients with T1-T3 esophageal cancer who received surgeries
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Radical resection of esophageal cancer

SUMMARY:
The real-world observational study was designed to explore lymph metastases and prognoses of the Chinese patients with thoracic T1-T3 esophageal cancer

DETAILED DESCRIPTION:
This trial is a real-world non-interventional observational study. The Chinese patients with thoracic T1-T3 esophageal cancer enrolled from Jan.1999 to Jun.2017 were included and the study data on pathologically diagnosed patient demographic/tumor biological characteristics were collected to evaluate the relevance of lymph metastases and prognoses of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old;
* Patients who received radical resection of esophageal cancer;
* Pathologically diagnosed patients with thoracic T1-T3 esophageal cancer after surgeries;

Exclusion Criteria:

* Patients who received upper gastrointestinal surgeries;
* Patients with second primary tumors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically diagnosed Chinese patients with thoracic T1-T3 esophageal cancer who received radical resection of esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 3673 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of lymph nodes and percentages of patients with surgeries | 1999 - 2017
  Numbers of lymph nodes and percentages of patients with surgeries in the patients with thoracic T1-T3 esophageal cancer

SECONDARY OUTCOMES:
Impact factors of lymph metastases | 1999 - 2017
  Impact factors of lymph metastases

OTHER OUTCOMES:
Effects of lymph metastases on overall survival | 1999 - 2017
  Effects on lymph metastases on overall survival in the patients with thoracic esophageal cancer
Effects of the numbers of lymph nodes on overall survival | 1999 - 2017
  Effects of the numbers of lymph nodes on overall survival in the patients with thoracic esophageal cancer who received lymphadenectomy
Effects of surgeries on the percentages of the patients with esophageal cancer who received lymphadenectomy | 1999 - 2017
  Effects of surgeries on the percentages of the thoracic T1-T3 patients with esophageal cancer who received lymphadenectomy
Effects of surgeries on the extents of the patients with esophageal cancer who received surgeries | 1999 - 2017
  Effects of surgeries on the extents of the thoracic T1-T3 patients with esophageal cancer who received surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Yin Li, Principal Investigator — Henan Cancer Hospital
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No